CLINICAL TRIAL: NCT05749406
Title: Parental Attitudes to Neoanus Dilatations Post-reconstruction in Anorectal Malformations
Acronym: PANDA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Verity Haffenden (Other)
Responsible Party: Sponsor-Investigator, Verity Haffenden, Clinical Research Fellow in Paediatric Surgery, Guy's and St Thomas' NHS Foundation Trust
Organization: Guy's and St Thomas' NHS Foundation Trust (Other)
Other Study IDs: 313255
Record Dates: First submitted 2022-12-13; First posted 2023-03-01 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-05

CONDITIONS: Anorectal Malformations
MeSH Terms: conditions — Anorectal Malformations | interventions — Focus Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Focus group — Small virtual focus group discussion about experiences/attitudes towards post-operative anal dilatation.
Other: Semi-structured interview — Individual virtual interview to ascertain participant's experiences of performing anal dilatation post-operatively for their child with an anorectal malformation.

SUMMARY:
The goal of this qualitative clinical trial is to learn about parental attitudes and experiences of performing post-operative dilatation anal dilatations for their child with an anorectal malformation. The main question it aims to answer are:

1. What are parental experiences/attitudes towards performing anal dilatations post-operatively.

In the first part of the study, participants will take part in a small virtual focus group discussion to identify themes to aid design of a semi-structured interview for part 2. In part 2, participants will undergo a virtual semi-structured interview. The answers will be recorded, anonymised, transcribed and undergo thematic analysis.

DETAILED DESCRIPTION:
Babies born without an anal opening require reconstructive surgery to create one, allowing them to pass stools. After the procedure, some surgeons recommend that parents perform routine dilatation of the anal opening using a metal rod dilator called a Hegar dilator. Recent studies have shown no difference in clinical outcomes for patients who have routine anal dilatation and those who do not. This study will look to find out the parental experiences and attitudes towards performing anal dilatation for their child.

The study will be formed of 2 parts. Participants will all be parents who were asked to perform routine anal dilatation post-operatively for their child born with an anorectal malformation. In part 1, a focus group will be conducted via Microsoft teams to ascertain themes to formulate the questions for part 2. In part 2, individual semi-structured interviews will be performed via MS teams. The interviews will be recorded, anonymised, transcribed and undergo analysis to assess for common themes.

The results will be published to guide professionals with regards to best practice and help inform parental discussions for new patients.

ELIGIBILITY:
Inclusion Criteria:

The parent of any patient who has:

* Undergone a posterior sagittal anorectoplasty for anorectal malformation and been recommended post-operative anal dilatations
* AND operation performed prior to November 2020
* AND able to understand and communicate in English
* AND with access to a mobile/computer with MS Teams

Exclusion Criteria:

The parent of any patient who had has:

* NOT undergone a posterior sagittal anorectoplasty for anorectal malformation
* AND/OR, NOT been recommended post-operative anal dilatations
* OR operated on after to November 2020
* OR unable to understand and communicate in English
* OR without access to a mobile/computer with access to MS Teams

Ages: 16 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parents of patients born with an anorectal malformation who have undergone anorectoplasty and been recommended post-operative anal dilatations.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Parental reported experience of anal dilatation | 3 months
  Parental reported experience of anal dilatation; This is a qualitative study that will use thematic analysis to identify parental reported experiences of performing anal dilatations in children. No scale/questionnaire will be used to allow for appropriate breadth of response.

IPD SHARING:
Plan to Share IPD: No
Patient data will not be shared at this stage